CLINICAL TRIAL: NCT02019693
Title: A Phase 2 Study of the MET Kinase Inhibitor INC280 in Papillary Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramaprasad Srinivasan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140037; 14-C-0037
Record Dates: First submitted 2013-12-20; First posted 2013-12-24 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Kidney Cancer
Keywords: Hereditary Papillary Renal Cell Carcinoma; VEGF Pathway; mTOR Inhibitor; Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Capmatinib (INC280) (Experimental): INC280 400 mg twice every day by mouth, continuously
  Interventions: Drug: INC280

INTERVENTIONS:
Drug: INC280 — Supplied by Novartis as film-coated tablet for oral use.
  Other Names: Capmatinib

SUMMARY:
Background:

* Papillary Renal Cell Cancer (RCC) is the second most common histologic subtype of kidney cancer, accounting for approximately 10-15% of cases
* Type 1 papillary RCC occurs in both sporadic and hereditary forms, which are histologically identical. Non familial type 1 papillary RCC can present as both solitary renal tumors and as bilateral, multifocal disease
* There are no standard agents of proven efficacy for patients with advanced papillary

RCC.

* Patients with disease localized to the kidney are managed surgically while patients with advanced/unresectable disease are usually managed in the community with vascular endothelial growth factor (VEGF) pathway antagonists or mechanistic target of rapamycin (mTOR) inhibitors.
* Activating mutations of mesenchymal epithelial transition (MET) were identified in the germline of affected hereditary papillary renal cancer (HPRC) patients, who have a predilection for the development of bilateral, multifocal type 1 papillary RCC. Somatic MET mutations have been found in a subset of patients with non-inherited, sporadic papillary renal carcinoma
* The investigational agent Capmatinib (INC280) is a selective MET inhibitor lacking activity against the VEGF pathway
* This is a proof-of-concept study using INC280 in patients with papillary RCC to test the idea that effectively blocking the hepatocyte growth factor (HGF)/MET pathway will lead to clinical activity in patients with papillary renal cell cancer

Objectives:

Primary Objective:

-To determine the overall response rate (Response Evaluation Criteria in Solid Tumors (RECIST) 1.1) in patients with papillary renal cell carcinoma treated with single agent INC280

Eligibility:

* Diagnosis of hereditary papillary renal carcinoma (HPRC) or sporadic papillary renal cell carcinoma (RCC)

  * Patients with bilateral multifocal disease can have tumors localized to the kidney or have metastatic disease
  * Patients with sporadic papillary RCC (but without multifocal disease) should have advanced disease that is considered unresectable
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Measurable disease
* Adequate organ function
* No active brain metastases
* Prior therapy

  * No more than 3 prior lines of systemic therapy
  * Prior therapy with a MET inhibitor is allowed as long as the patient has not had progressive disease while receiving the agent

Design:

* This is a phase 2 single center non-randomized trial.
* The study will be conducted using a Simon 2 stage minimax design. Initially 13 evaluable subjects will be recruited. If there are no responses to therapy, the study will be terminated. If there is at least 1 response an additional 7 evaluable subjects will be accrued.
* The two-stage minimax design is based on assuming an ineffective response rate of 5% and a targeted effective response rate of 25%. We also assume that the probability of accepting an ineffective treatment and the probability of rejecting an effective treatment are each 10%.
* Subjects will be dosed orally at a starting dose of 600 mg twice daily.
* The overall response rate (complete response + partial response) will be determined.

DETAILED DESCRIPTION:
Background:

* Papillary Renal Cell Cancer (RCC) is the second most common histologic subtype of kidney cancer, accounting for approximately 10-15% of cases
* Type 1 papillary RCC occurs in both sporadic and hereditary forms, which are histologically identical. Non familial type 1 papillary RCC can present as both solitary renal tumors and as bilateral, multifocal disease
* There are no standard agents of proven efficacy for patients with advanced papillary

RCC.

* Patients with disease localized to the kidney are managed surgically while patients with advanced/unresectable disease are usually managed in the community with vascular endothelial growth factor (VEGF) pathway antagonists or mechanistic target of rapamycin (mTOR) inhibitors.
* Activating mutations of mesenchymal epithelial transition (MET) were identified in the germline of affected HPRC patients, who have a predilection for the development of bilateral, multifocal type 1 papillary RCC. Somatic MET mutations have been found in a subset of patients with non-inherited, sporadic papillary renal carcinoma
* The investigational agent Capmatinib (INC280) is a selective MET inhibitor lacking activity against the VEGF pathway
* This is a proof-of-concept study using INC280 in patients with papillary RCC to test the idea that effectively blocking the hepatocyte growth factor (HGF)//MET pathway will lead to clinical activity in patients with papillary renal cell cancer

Objectives:

Primary Objective:

-To determine the overall response rate (Response Evaluation Criteria in Solid Tumors (RECIST) 1.1) in patients with papillary renal cell carcinoma treated with single agent INC280

Eligibility:

* Diagnosis of hereditary papillary renal carcinoma (HPRC) or sporadic papillary renal cell carcinoma (RCC)

  * Patients with bilateral multifocal disease can have tumors localized to the kidney or have metastatic disease
  * Patients with sporadic papillary RCC (but without multifocal disease) should have advanced disease that is considered unresectable
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Measurable disease
* Adequate organ function
* No active brain metastases
* Prior therapy

  * No more than 3 prior lines of systemic therapy
  * Prior therapy with a MET inhibitor is allowed as long as the patient has not had progressive disease while receiving the agent

Design:

* This is a phase 2 single center non-randomized trial.
* The study will be conducted using a Simon 2 stage minimax design. Initially 13 evaluable subjects will be recruited. If there are no responses to therapy, the study will be terminated. If there is at least 1 response an additional 7 evaluable subjects will be accrued.
* The two-stage minimax design is based on assuming an ineffective response rate of 5% and a targeted effective response rate of 25%. We also assume that the probability of accepting an ineffective treatment and the probability of rejecting an effective treatment are each 10%.
* Subjects will be dosed orally at a starting dose of 400 mg twice daily.
* The overall response rate (complete response + partial response) will be determined.

ELIGIBILITY:
* INCLUSION CRITERIA

2.1.1.1 Patients must have histologically or cytologically confirmed papillary Renal Cell Cancer (RCC).

1. Patients with bilateral multifocal disease can have tumors localized to the kidney or have metastatic disease
2. Patients with sporadic papillary RCC (but without multifocal disease) should have advanced disease that is considered unresectable

2.1.1.2 Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions). Nodal lesions must be 15mm by computed tomography (CT) scan or magnetic resonance imaging (MRI). Non nodal lesions must be >10 mm with CT scan or MRI.

2.1.1.3 Patients must have normal organ and marrow function as defined below:

* Hemoglobin > 9 g/dL (SI Units: 90 g/L)
* Platelet count greater than or equal to 75 x 10 (9)/L
* Absolute neutrophil count (ANC) greater than or equal to 1.5 x 10(9)/L without growth factor support
* Total bilirubin less than or equal to 2 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and/or alanine aminotransferase (ALT)/serum glutamate-pyruvate transaminase (SGPT) less than or equal to 2.5 x upper limit of normal (ULN)
* Serum creatinine less than or equal to 1.5 x ULN
* Asymptomatic serum amylase less than or equal to 2 x ULN; patients with > ULN but less than or equal to 2 x ULN serum amylase at study start must be confirmed to have no signs and/or symptoms suggestion pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
* Serum lipase less than or equal to ULN
* Fasting serum triglyceride level less than or equal to 500 mg/dL

2.1.1.4 Patients may have had no more than 3 prior lines of systemic therapy. Prior therapy with a mesenchymal epithelial transition (MET) inhibitor is allowed as long as the patient has not had progressive disease while receiving the agent

2.1.1.5 Patient must be able to swallow and retain oral medication

2.1.1.6 Age greater than or equal to18 years.

2.1.1.7 Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.

2.1.1.8 Patients must provide written informed consent prior to any study procedures.

2.1.1.9 Patients must be willing and able to comply with scheduled visits, treatment plan and laboratory tests

EXCLUSION CRITERIA

2.1.2.1 Patients who are receiving any other investigational agents for treatment of their kidney cancer.

2.1.2.2 History of allergic reactions attributed to compounds of similar chemical or biologic composition to Capmatinib (INC280). Excipients in the current formulation include microcrystalline cellulose, mannitol, sodium starch glycolate, magnesium stearate and colloidal silicon dioxide

2.1.2.3 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or potentially affect the interpretation of study data.

2.1.2.4 Subjects with significant or uncontrolled cardiovascular disease (e.g., uncontrolled hypertension, peripheral vascular disease, congestive heart failure, cardiac arrhythmia, or acute coronary syndrome) within 6 months prior to starting study treatment or heart attack within 12 months prior to starting study treatment

2.1.2.5 Patients receiving any medications that are known to be strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4), or sensitive substrates of CYP3A4, cytochrome P450 1A2 (CYP1A2), cytochrome P450 family 2 subfamily C member 9 (CYP2C9), cytochrome P450 2C19 (CYP2C19) or P-glycoprotein (P-gp) with a narrow therapeutic index.

2.1.2.6 Symptomatic central nervous system (CNS) metastases that are neurologically unstable or requiring > 5 mg/day of dexamethasone (or equivalent) to control CNS disease.

Note: Patients with controlled CNS metastases are allowed. Radiotherapy or surgery for CNS metastases must have been completed >2 weeks prior to study entry. Patients must be neurologically stable, having no new neurologic deficits on clinical examination, and no new findings on CNS imaging. Steroid use for management of CNS metastases must be at a stable dose for two weeks preceding study entry.

2.1.2.7 Patients with greater than or equal to Grade 2 neuropathy.

2.1.2.8 Treatment with proton pump inhibitors within 3 days prior to study entry. If continued use of gastrointestinal (GI) prophylaxis is required, the patient will be switched to an appropriate Histamine H2-receptor antagonists (H2) with appropriate counsel and caution.

2.1.2.9 Currently receiving any prohibited medications including vitamins and herbal Supplements.

2.1.2.10 Major surgery within 4 weeks prior to initiating treatment, excluding the placement of vascular access.

2.1.2.11 The subject has not recovered to baseline, Common Terminology Criteria for Adverse Events (CTCAE) less than or equal to Grade 1 from toxicity due to all prior therapies for RCC or to a level permitted under other sections of the eligibility criteria except alopecia and other non-clinically significant adverse events (AEs).

2.1.2.12 Any other condition that would, in the Investigators judgment, contraindicate participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.

2.1.2.13 Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 30 mIU/mL). Laboratory values >5 mIU/mL, but <30 mIU/mL should be repeated in 48 hours.

2.1.2.14 Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months days after stopping study drug. Highly effective contraception methods include:

* Total abstinence or
* Male or female sterilization or
* Combination of any two of the following (a+b or a+c or b+c):

  1. Use of oral, injected or implanted hormonal methods of contraception
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

2.1.2.15 Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

2.1.2.16 Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Capmatinib (INC280).

2.1.2.17 Prior invasive malignancy of other histology currently requiring treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaprasad Srinivasan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0037.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Capmatinib (INC280): Participants received a starting dose of 600mg twice a day (BID) of capmatinib initially; following a change in formulation during the study, the starting dose was changed to 400mg BID, based on pharmacokinetic (PK) studies that demonstrated that this corresponded to the starting dose of 600mg BID of the old formulation.
Period: Overall Study
Arm/Group | Capmatinib (INC280)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.63 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions. Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From start of study until permanent treatment discontinuation (range 2 weeks-238 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
percentage of participants
  Complete Response | 0
  Partial Response | 15
  Stable Disease | 65
  Progressive Disease | 10
  Not evaluable for response | 10

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: Median 26.8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Months | 10.2 [3.67 to NA] — The upper bounds of the 95% confidence interval (CI) were not reached at the time of this analysis.

3. Secondary Outcome: Overall Survival
Description: OS is the time between the first day of treatment and day of death or last follow up calculated by Kaplan Meier analysis.
Time Frame: Median 26.8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Months | 31 [21.9 to NA] — The upper bounds of the 95% confidence interval (CI) were not reached at the time of this analysis.

4. Secondary Outcome: Disease Control Rate (Partial and Complete Response Plus Stable Disease > 6 Months)
Description: Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is disappearance of all target lesions. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From start of study until permanent treatment discontinuation (range 2 weeks-238 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
percentage of participants | 35

5. Secondary Outcome: Number of Grades 1-5 Adverse Events Related to Treatment
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 94 months and 21 days
Measure: Number; unit: adverse events
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
adverse events
  Grade 1 | 228
  Grade 2 | 81
  Grade 3 | 13
  Grade 4 | 3
  Grade 5 | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 94 months and 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Capmatinib (INC280)
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 94 months and 21 days.
Arm/Group | Capmatinib (INC280)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capmatinib (INC280) (N=20)
Alanine aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Thyroid mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pain (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capmatinib (INC280) (N=20)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Alanine aminotransferase increased (Investigations) | 5 (10)
Alkaline phosphatase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (13)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (7)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 1 (1)
CPK increased (Investigations) | 2 (14)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 6 (7)
Cholesterol high (Investigations) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Creatinine increased (Investigations) | 15 (49)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (19)
Dizziness (Nervous system disorders) | 6 (9)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 12 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema face (General disorders) | 1 (2)
Edema limbs (General disorders) | 9 (32)
Eye disorders - Other, Left eye subconjunctival hemorrhage (Eye disorders) | 1 (1)
Eye disorders - Other, Right eye stye (Eye disorders) | 1 (1)
Fatigue (General disorders) | 11 (17)
Fever (General disorders) | 4 (6)
Flashing lights (Eye disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other, diverticulosis (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Sweats (General disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 2 (6)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (8)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (14)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 2 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (19)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (7)
Hyponatremia (Metabolism and nutrition disorders) | 6 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (21)
Hypotension (Vascular disorders) | 5 (6)
Hypothyroidism (Endocrine disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Irritability (General disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increased (Investigations) | 7 (16)
Localized edema (General disorders) | 1 (4)
Lymphocyte count decreased (Investigations) | 11 (27)
Memory impairment (Nervous system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Nausea (Gastrointestinal disorders) | 16 (20)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Benign Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders - Other, numbness sinus area (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (28)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 10 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 6 (18)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Serum amylase increased (Investigations) | 6 (9)
Sinus bradycardia (Cardiac disorders) | 5 (11)
Skin and subcutaneous tissue disorders - Other, Seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (10)
Weight gain (Investigations) | 4 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT02019693/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT02019693/ICF_001.pdf